CLINICAL TRIAL: NCT00508898
Title: The Efficacy and Safety of Calcitriol for the Treatment of Lupus Nephritis and Persistent Proteinuria
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding problem; trial abandoned.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: SZETO, Cheuk Chun, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2007.261-T
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2009-01

CONDITIONS: Systemic Lupus Erythematosus; Nephritis; Proteinuria
Keywords: lupus nephritis; proteinuria; chronic kidney diseases; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Nephritis; Proteinuria; Lupus Nephritis; Renal Insufficiency, Chronic | interventions — Calcitriol; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment group (Experimental): Patients will receive calcitriol at a fixed dose of 1 mcg twice weekly.
  Interventions: Drug: Calcitriol
- control group (Active Comparator): Patients will receive multivitamin 1 tab daily (with vitamin D2 300 IU).
  Interventions: Drug: Multivitamin

INTERVENTIONS:
Drug: Calcitriol — Patients will receive calcitriol (oral capsule) at a fixed dose of 1 mcg twice weekly.
  Arms: treatment group
Drug: Multivitamin — Patients will receive multivitamin 1 tab daily (with vitamin D2 300 IU).
  Arms: control group

SUMMARY:
Glomerulonephritis and renal failure represent one of the most life-threatening manifestations of systemic lupus erythematosus (SLE). Although immunosuppressive therapy is often effective for the treatment of acute lupus nephritis, a significant proportion of patients show persistent proteinuria after resolution of the acute nephritic process, and develop progressive renal failure. There is preliminary evidence that calcitriol and other vitamin D analogs can reduce proteinuria in patients with chronic kidney diseases. The investigators plan to conduct a randomized control study to evaluate the safety and efficacy of calcitriol in the treatment of SLE patients with persistent proteinuria. Sixty patients with clinically quiescent SLE and persistent proteinuria despite conventional therapy will be recruited. They will be treated with calcitriol for 48 weeks. Proteinuria, renal function, lupus disease activity, serum and urinary inflammatory markers will be monitored. This study will explore the potential anti-proteinuric and immunomodulating effects of calcitriol in the treatment of SLE, which is a common and life threatening disease in young adults.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* clinical quiescent SLE for at least 12 weeks
* baseline SLEDAI score <= 4
* history of biopsy-proven lupus nephritis
* estimated glomerular filtration rate 15 to 60 ml/min/1.73m2
* proteinuria > 1 g/day (or proteinuria > 1 g/g-Cr) in 2 consecutive samples within 12 weeks despite ACE inhibitor or angiotensin receptor blocker for at least 3 months
* on maintenance dose of prednisolone < 10 mg/day, with or without other immunosuppressive medications
* corrected serum calcium level < 2.45 mmol/l
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* History of malignancy, including leukemia and lymphoma within the past 2 years
* Systemic infection requiring therapy at study entry
* Any other severe coexisting disease such as, but not limited to, chronic liver disease, myocardial infarction, cerebrovascular accident, malignant hypertension
* History of drug or alcohol abuse within past 2 years
* Participation in any previous trial on vitamin D analogue
* Patients receiving treatment of vitamin D and/or its analogue for other medical reasons within the past 4 weeks. Patients who are taking multivitamin supplement that contains vitamin D could be enrolled after 4 weeks of wash out period by changing to a preparation that has no vitamin D.
* On other investigational drugs within last 30 days
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance
* Known history of sensitivity or allergy to vitamin D analogs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
change in proteinuria | one year

SECONDARY OUTCOMES:
Secondary end points include risk of lupus flare, change in renal function, Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score, serum and urinary inflammatory markers. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk-Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong